CLINICAL TRIAL: NCT00866658
Title: A Randomized, Double-Blind, Placebo-Controlled, 2-arm Parallel-group, Multicenter Study With a 24-Week Treatment Period Assessing the Efficacy and Safety of AVE0010 in Patients With Type 2 Diabetes Insufficiently Controlled With Basal Insulin With or Without Sulfonylurea
Brief Title: GLP-1 Receptor Agonist Lixisenatide in Patients With Type 2 Diabetes for Glycemic Control and Safety Evaluation, on Top of Basal Insulin +/- Sulfonylurea (GETGOAL-L-ASIA)
Acronym: GETGOAL-L-ASIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC10887
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: hyperglycemia; GLP-1; sulfonylurea; insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Insulin Resistance | interventions — lixisenatide; Sulfonylurea Compounds

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lixisenatide (Experimental): 2-step initiation regimen of lixisenatide: 10 microgram (mcg) once daily (QD) for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to Week 24.
  Interventions: Drug: Lixisenatide (AVE0010); Device: Pen auto-injector; Drug: Sulfonylurea; Drug: Basal Insulin
- Placebo (Placebo Comparator): 2-step initiation regimen of volume matching placebo: 10 mcg QD for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to Week 24.
  Interventions: Drug: Placebo; Device: Pen auto-injector; Drug: Sulfonylurea; Drug: Basal Insulin

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Self-administered by subcutaneous injections once daily within the hour preceding breakfast.
  Arms: Lixisenatide
Drug: Placebo — Self-administered by subcutaneous injections once daily within the hour preceding breakfast.
  Arms: Placebo
Device: Pen auto-injector
  Other Names: OptiClik®
Drug: Sulfonylurea — Sulfonylurea if given, to be continued at a stable dose.
Drug: Basal Insulin — To be continued at a stable dose.

SUMMARY:
The purpose of this study is to evaluate the benefits and risks of lixisenatide (AVE0010), in comparison to placebo, as an add-on treatment to basal insulin with or without sulfonylurea, over a period of 24 weeks of treatment.

The primary objective is to assess the effects of lixisenatide, when added to basal insulin, on glycemic control in terms of glycosylated hemoglobin (HbA1c) reduction at Week 24.

The secondary objectives are to assess the effects of lixisenatide on body weight, 2-hour postprandial plasma glucose (PPG) after standardized meal challenge test, percentage of patients reaching HbA1c less than 7 percent (%), percentage of patients reaching HbA1c less than or equal to 6.5%, fasting plasma glucose (FPG), change in 7-point self-monitored plasma glucose (SMPG) profiles, change in daily basal insulin and total insulin doses; to evaluate safety, tolerability, pharmacokinetics (PK), and anti-lixisenatide antibody development.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus, diagnosed for at least 1 year at the time of the screening visit, insufficiently controlled with basal insulin with or without sulfonylurea

Exclusion Criteria:

* HbA1c less than (<) 7 percent (%) or greater than (>) 10% at screening
* At the time of screening age <legal age of majority
* Pregnant or breastfeeding women or women of childbearing potential with no effective contraceptive method
* Type 1 diabetes mellitus
* Treatment with basal insulin for less than 3 months prior to screening or insulin regimen changed during the last 3 months prior to screening
* Basal insulin dose at screening <10 units/day and/or during the last 2 months dose not stable (+/- 20%)
* Sulfonylurea not at a stable (unchanged) dose for at least 3 months prior to screening
* FPG at screening >250 milligram/deciliter (mg/dL) (>13.9 millimole/liter [mmol/L])
* History of hypoglycemia unawareness
* Weight change of more than 5 kilogram (kg) during the 3 months preceding the screening visit
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery, inflammatory bowel disease
* History of metabolic acidosis, including diabetic ketoacidosis within 1 year prior to screening
* Hemoglobinopathy or hemolytic anemia, receipt of blood or plasma products within 3 months prior to the time of screening
* Within the last 6 months prior to screening: history of myocardial infarction, stroke, or heart failure requiring hospitalization
* Known history of drug or alcohol abuse within 6 months prior to the time of screening
* Cardiovascular, hepatic, neurological, endocrine disease, active malignant tumor or other major systemic disease or patients with short life expectancy making implementation of the protocol or interpretation of the study results difficult, history or presence of clinically significant diabetic retinopathy, history or presence of macular edema likely to require laser treatment within the study period
* Uncontrolled or inadequately controlled hypertension at the time of screening with a resting systolic blood pressure or diastolic blood pressure >180 millimeter of mercury (mmHg) or >95 mmHg, respectively
* Laboratory findings at the time of screening: aspartate aminotransferase, alanine aminotransferase, or alkaline phosphatase: >2 times upper limit of the normal (ULN) laboratory range; amylase and/or lipase: >3 times ULN; total bilirubin: >1.5 times ULN (except in case of Gilbert's syndrome); hemoglobin <11 gram/deciliter and/or neutrophils <1500 per cubic millimeter (mm^3) and/or platelets <100 000/mm^3; positive test for Hepatitis B surface antigen and/or Hepatitis C antibody and positive serum pregnancy test in females of childbearing potential
* Any clinically significant abnormality identified on physical examination, laboratory tests, electrocardiogram, or vital signs at the time of screening that, in the judgment of the investigator or any sub-investigator, precludes safe completion of the study or constrains efficacy assessment
* Patients who are considered by the investigator as inappropriate for this study for any reason (for example, impossibility to meet specific protocol requirements, such as scheduled visits, being able to do self-injections, likelihood of requiring treatment during the screening phase and treatment phase with drugs not permitted by the clinical study protocol)
* Patient was an investigator or any sub-investigator, pharmacist, study coordinator, other study staff or relative thereof directly involved in the conduct of the protocol
* Use of other oral or injectable antidiabetic or hypoglycemic agents other than sulfonylurea or basal insulin (for example, metformin, alpha glucosidase inhibitor, thiazolidinedione, rimonabant, exenatide, dipeptidyl peptidase 4 inhibitors, fast acting insulin for 1 week or more etc.) within 3 months prior to the time of screening
* Use of systemic glucocorticoids (excluding topical application or inhaled forms) for 1 week or more within 3 months prior to the time of screening
* Use of any investigational drug within 3 months prior to screening
* Participation in any previous study with lixisenatide
* End-stage renal disease defined by a serum creatinine clearance of <15 milliliter/minute (mL/min) (calculated by the Cockcroft and Gault formula) and/or patients on dialysis
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including, but not limited to gastroparesis and gastroesophageal reflux disease requiring medical treatment, within 6 months prior to the time of screening
* Allergic reaction to any glucagon like peptide-1 (GLP-1) agonist in the past (for example, exenatide, liraglutide) or to metacresol
* Additional exclusion criteria at the end of the run-in phase: informed consent withdrawal; lack of compliance during the single-blind placebo run-in phase (>2 injections missed); and patient with any adverse event which could have precludes the inclusion in the study, as assessed by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- Sanofi-Aventis Administrative Office, Tokyo, Japan
- Sanofi-Aventis Administrative Office, Makati City, Philippines
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Taipei, Taiwan

REFERENCES:
- [Result] Seino Y, Min KW, Niemoeller E, Takami A; EFC10887 GETGOAL-L Asia Study Investigators. Randomized, double-blind, placebo-controlled trial of the once-daily GLP-1 receptor agonist lixisenatide in Asian patients with type 2 diabetes insufficiently controlled on basal insulin with or without a sulfonylurea (GetGoal-L-Asia). Diabetes Obes Metab. 2012 Oct;14(10):910-7. doi: 10.1111/j.1463-1326.2012.01618.x. Epub 2012 May 30. PMID 22564709
- [Derived] Davidson JA, Stager W, Paranjape S, Berria R, Leiter LA. Achieving postprandial glucose control with lixisenatide improves glycemic control in patients with type 2 diabetes on basal insulin: a post-hoc analysis of pooled data. Clin Diabetes Endocrinol. 2020 Jan 14;6:2. doi: 10.1186/s40842-019-0088-5. eCollection 2020. PMID 31956422
- [Derived] Seino Y, Ikeda Y, Niemoeller E, Watanabe D, Takagi H, Yabe D, Inagaki N. Efficacy and Safety of Lixisenatide in Japanese Patients with Type 2 Diabetes Insufficiently Controlled with Basal Insulin+/-Sulfonylurea: A Subanalysis of the GetGoal-L-Asia Study. Horm Metab Res. 2015 Nov;47(12):895-900. doi: 10.1055/s-0035-1549875. Epub 2015 Jun 3. PMID 26039935

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 57 centers in 4 countries between March 10, 2009 and June 23, 2010.
Pre-assignment Details: A total of 437 patients were screened of which 126 (28.8%) were screen failures; main reason for screen failure was glycosylated hemoglobin (HbA1c) values being out of the defined protocol range (greater than or equal to 7% and less than or equal to 10%). A total of 311 patients were randomized.
Groups:
- Placebo: 2-step initiation regimen of volume matching placebo: 10 microgram (mcg) once daily (QD) subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to Week 24.
- Lixisenatide: 2-step initiation regimen of lixisenatide: 10 mcg QD subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to Week 24.
Period: Overall Study
Arm/Group | Placebo | Lixisenatide
Started | 157 (Randomized.) | 154
Safety Population | 157 (All patients who were exposed to at least 1 dose, regardless of amount of treatment administered.) | 154
Modified Intent-to-Treat(mITT)Population | 157 (All patients who received at least 1 dose;had baseline,at least 1 post-baseline efficacy assessment.) | 154
Completed | 144 | 133
Not Completed | 13 | 21
Not completed — Adverse Event | 5 | 14
Not completed — Lack of Efficacy | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Familial and Personal Reasons | 4 | 5

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Groups:
- Placebo: 2-step initiation regimen of volume matching placebo: 10 mcg QD subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to Week 24.
- Total: Total of all reporting groups
Arm/Group | Placebo | Lixisenatide | Total
Number analyzed (Participants) | 157 | 154 | 311
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (10.1) | 58.7 (10.2) | 58.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 85 | 162
  Male | 80 | 69 | 149
Race/Ethnicity, Customized [Number; unit: participants]
  Race: Asian/Oriental | 157 | 154 | 311
  Ethnicity: Non Hispanic | 157 | 154 | 311
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of hemoglobin] | 8.52 (0.78) | 8.54 (0.73) | 8.53 (0.76)
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 65.60 (12.47) | 65.93 (13.00) | 65.77 (12.72)
2-Hour Postprandial Plasma Glucose (PPG) [Mean (Standard Deviation); unit: millimole per liter (mmol/L)] — The 2-hour PPG test measured blood glucose 2 hours after eating a standardized meal. Number of patients analyzed = 156 and 152 for Placebo and Lixisenatide treatment arms, respectively.
  millimole per liter (mmol/L) | 17.75 (3.94) | 17.81 (3.36) | 17.78 (3.66)
Number of Patients With Screening HbA1c Less Than 8% [Number; unit: participants] | 36 | 35 | 71
Number of Patients With Screening HbA1c Greater Than or Equal to 8% [Number; unit: participants] | 121 | 119 | 240
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 7.75 (2.25) | 7.67 (2.32) | 7.71 (2.28)
Average 7-point Self-Monitored Plasma Glucose (SMPG) [Mean (Standard Deviation); unit: mmol/L] — Here, number of patients analyzed = 139 and 147 for Placebo and Lixisenatide treatment arms, respectively.
  mmol/L | 11.42 (2.46) | 11.58 (2.51) | 11.51 (2.48)
Glucose Excursion [Mean (Standard Deviation); unit: mmol/L] — Glucose excursion = 2-hour PPG minus plasma glucose 30 minutes prior to the meal test, before study drug administration. Number of patients analyzed = 156 and 152 for Placebo and Lixisenatide treatment arms, respectively.
  mmol/L | 9.70 (4.19) | 9.72 (3.27) | 9.71 (3.75)
Basal Insulin Treatment Duration [Mean (Standard Deviation); unit: years] — Basal insulin treatment duration is reported at screening. Number of patients analyzed = 155 and 154 for Placebo and Lixisenatide treatment arms, respectively.
  years | 3.01 (4.27) | 2.94 (3.67) | 2.97 (3.97)
Total Insulin Dose [Mean (Standard Deviation); unit: units per day] — Total insulin dose is reported at screening.
  units per day | 24.11 (14.18) | 24.85 (13.96) | 24.48 (14.05)
Number of Patients With Insulin Therapy at Screening [Number; unit: participants] — NPH included isophane insulin and insulin human injection, isophane. Premix insulin included Novomix.
  participants
    Glargine | 92 | 95 | 187
    Detemir | 42 | 41 | 83
    Neutral Protamine Hagedorn (NPH) | 21 | 18 | 39
    Premix (Mixed Insulin) | 2 | 0 | 2
Duration of Diabetes [Mean (Standard Deviation); unit: years] — Duration of diabetes is reported at screening.
  years | 14.13 (7.72) | 13.71 (7.73) | 13.92 (7.71)
Sulfonylurea Treatment Duration [Mean (Standard Deviation); unit: years] — Sulfonylurea treatment duration is reported at screening. Number of patients analyzed = 101 and 100 for Placebo and Lixisenatide treatment arms, respectively.
  years | 6.80 (5.24) | 5.33 (4.83) | 6.07 (5.08)
Number of Patients With Sulfonylurea Use [Number; unit: participants] — Number of patients with sulfonylurea urea is reported at screening.
  participants
    Yes | 111 | 108 | 219
    No | 46 | 46 | 92
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — Body mass index was calculated by dividing body weight (kilogram) by the height (meters) squared.
  kilogram per square meter (kg/m^2) | 25.15 (3.94) | 25.36 (3.69) | 25.26 (3.82)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 3 days after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population:all randomized patients who received at least 1 dose;had baseline,at least 1 post-baseline efficacy assessment, irrespective of compliance with study protocol/procedures. Last observation carried forward used. Number of patients analyzed=patients with baseline and at least 1 post-baseline HbA1c assessment during on treatment period.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Groups:
- Placebo: 2-step initiation regimen up to a maintenance dose of 20 mcg of volume matching placebo.
- Lixisenatide: 2-step initiation regimen up to a maintenance dose of 20 mcg of lixisenatide.
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 154 | 146
percentage of hemoglobin | 0.11 (0.131) | -0.77 (0.137)
Statistical Analysis 1: Comparison: Placebo vs Lixisenatide; To detect a difference of 0.5% in change from baseline to Week 24 in HbA1c between lixisenatide and placebo, 145 patients in each arm would provide a power of 90% assuming common standard deviation of 1.3% with a 2-sided t test at 5% significance level; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing: 2-sided at significance level=0.05. Analysis of co-variance(ANCOVA)included treatment arms, randomization strata of screening HbA1c (<8.0, >=8.0%),sulfonylurea use (yes, no), country as fixed effects, baseline HbA1c as covariate; Least squares (LS) mean difference = -0.88, 95% CI 2-sided [-1.116 to -0.650], Standard Error of Mean 0.118

2. Secondary Outcome: Change From Baseline in 2-hour Postprandial Plasma Glucose (PPG) at Week 24
Description: The 2-hour PPG test measured blood glucose 2 hours after eating a standardized meal. Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to the last dosing day of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using last observation carried forward (LOCF). Here, number of patients analyzed = patients with baseline and at least 1 post-baseline 2-hour PPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 142 | 131
mmol/L | -0.14 (0.563) | -7.96 (0.598)

3. Secondary Outcome: Change From Baseline in Body Weight at Week 24
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline body weight assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 157 | 150
kilogram | 0.06 (0.271) | -0.38 (0.284)

4. Secondary Outcome: Change From Baseline in Average 7-Point Self Monitored Plasma Glucose (SMPG) Profile at Week 24
Description: Patients recorded a 7-point plasma glucose profile measured before and 2 hours after each meal and at bedtime once in a week and the average value for the 7-time points was calculated. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to the last dosing day of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline average 7-point SMPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 138 | 142
mmol/L | -0.56 (0.271) | -1.91 (0.272)

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 1 day after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline FPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 157 | 148
mmol/L | 0.25 (0.302) | -0.42 (0.314)

6. Secondary Outcome: Change From Screening in Total Insulin Dose at Week 24
Description: Change was calculated by subtracting screening value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to the last dosing day of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Screening, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post baseline insulin dose assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: units per day
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 157 | 151
units per day | -0.11 (0.442) | -1.39 (0.458)

7. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than 7% at Week 24
Description: The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 3 days after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 154 | 146
percentage of participants | 5.2 | 35.6

8. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than or Equal to 6.5% at Week 24
Description: as for outcome 7
Time Frame: Week 24
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 154 | 146
percentage of participants | 1.3 | 17.8

9. Other Pre Specified Outcome: Change From Baseline in Glucose Excursion at Week 24
Description: Glucose excursion = 2-hour PPG minus plasma glucose 30 minutes prior to the standardized meal test, before study drug administration. Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to the last dosing day of the study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline glucose excursion assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 142 | 131
mmol/L | 0.14 (0.542) | -7.09 (0.576)

10. Other Pre Specified Outcome: Percentage of Patients With at Least 5% Weight Loss From Baseline at Week 24
Description: as for outcome 7
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 157 | 150
percentage of participants | 4.5 | 7.3

11. Secondary Outcome: Percentage of Patients Requiring Rescue Therapy During 24-Week Period
Description: Routine fasting SMPG and central laboratory FPG (and HbA1c after week 12) values were used to determine the requirement of rescue medication. If fasting SMPG value exceeded the specified limit for 3 consecutive days, the central laboratory FPG (and HbA1c after week 12) were performed. Threshold values - from baseline to Week 8: fasting SMPG/FPG >270 milligram/deciliter (mg/dL) (15.0 mmol/L), from Week 8 to Week 12: fasting SMPG/FPG >240 mg/dL (13.3 mmol/L), and from Week 12 to Week 24: fasting SMPG/FPG >200 mg/dL (11.1 mmol/L) or HbA1c >8.5%. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline up to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 157 | 154
percentage of participants | 3.2 | 1.3

12. Other Pre Specified Outcome: Number of Patients With Symptomatic Hypoglycemia and Severe Symptomatic Hypoglycemia
Description: Symptomatic hypoglycemia was an event with clinical symptoms that were considered to result from a hypoglycemic episode with an accompanying plasma glucose less than 60 mg/dL (3.3 mmol/L) or associated with prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration if no plasma glucose measurement was available. Severe symptomatic hypoglycemia was symptomatic hypoglycemia event in which the patient required the assistance of another person and was associated with either a plasma glucose less than 36 mg/dL (2.0 mmol/L) or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration, if no plasma glucose measurement was available.
Time Frame: First dose of study drug up to 3 days after the last dose administration
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 157 | 154
participants
  Symptomatic hypoglycemia | 37 | 66
  Severe symptomatic hypoglycemia | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 3 days after the last dose administration
Description: Median exposure to study treatment was 169 days in both arms. The analysis was performed on safety population, defined as all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Arm/Group | Placebo | Lixisenatide
Serious Adverse Events (participants affected / at risk) | 9/157 | 10/154
Other Adverse Events (participants affected / at risk) | 71/157 | 125/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=157) | Lixisenatide (N=154)
Herpes zoster oticus (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 2
Hyphaema (Eye disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=157) | Lixisenatide (N=154)
Nasopharyngitis (Infections and infestations) | 20 | 21
Decreased appetite (Metabolism and nutrition disorders) | 0 | 10
Hypoglycaemia (Metabolism and nutrition disorders) | 37 | 67 — Hypoglycaemia adverse event is based on investigator reported hypoglycaemia.
Dizziness (Nervous system disorders) | 8 | 13
Headache (Nervous system disorders) | 3 | 16
Abdominal discomfort (Gastrointestinal disorders) | 1 | 11
Constipation (Gastrointestinal disorders) | 4 | 8
Diarrhoea (Gastrointestinal disorders) | 4 | 10
Dyspepsia (Gastrointestinal disorders) | 0 | 11
Nausea (Gastrointestinal disorders) | 7 | 61
Vomiting (Gastrointestinal disorders) | 3 | 28
Asthenia (General disorders) | 12 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.